CLINICAL TRIAL: NCT07250490
Title: Cross-Cultural Adaptation to Portuguese and Psychometric Validation of the DIVA Questionnaire (Day-to-Day Impact of Vaginal Aging)
Brief Title: Validation of the DIVA (Day to Day Impact of Vaginal Aging) Questionnaire for Portuguese Women
Status: Completed | Type: Observational
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Hospital Santo André - Centro Hospitalar de Leiria (Unknown); University of Minho (Other)
Responsible Party: Principal Investigator, AndreiaAntunes, affiliated investigator, PhD Student, Consultant of Gynecology and Obstetrics, Instituto Politécnico de Leiria
Other Study IDs: 6047/2022 CES ARS-LVT
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Vulvovaginal Atrophy; Genital Disorder; PROMs
Keywords: Genitourinary syndrome of menopause (GSM); Female Genital Atrophy; Female Sexual Dysfunction (FSD); Dyspareunia; Female Genital Disorder; Vaginal dryness; Vaginal Itching
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult women attending a clinical appointment: Adult women attending medical appointments. For the convenience normative sample of the general population will include users of a health center large urban healthcare; the Personalized Health Care Unit (UCSP) of Sete Rios, in Lisbon. For the convenience clinical sample, users of the general gynecology consultation at a private hospital (Hospital Dom Manuel de Aguiar) and the gynecology consultation at a public hospital (Hospital Santo André), units located in an urban center in Leiria. Those from a private clinic in the north of the country, in Braga, will also be included. It is intended to include a minimum of 230 questionnaires, according to the recommendation of the COSMIN13, to allow an assessment of invariance correlation

SUMMARY:
To determine the reliability and validity of the Portuguese version of the DIVA questionnaire in Portuguese women. This validation will support its use both in research and in routine clinical practice in this population.

DETAILED DESCRIPTION:
Prior to the initiation of this research protocol, the DIVA questionnaire was translated into European Portuguese following recommended best-practice guidelines. The process included the following sequential steps: (1) forward translation by two independent investigators; (2) reconciliation of the translations; (3) back-translation by two certified translators fluent in English; (4) unification and harmonization of the Portuguese version; (5) expert review by a panel of specialists in gynecology and sexology; and (6) pretesting in a group of patients, with final cultural adaptation of the DIVA scale into European Portuguese.

Symptoms that cannot be directly quantified but significantly affect quality of life can be assessed through self-reported health questionnaires. These clinical instruments play a key role: not only in identifying the clinical problem, but also in evaluating its individual impact across multiple psychological and physical dimensions, thereby helping to determine the effectiveness of therapeutic strategies in improving such subjective symptoms. For research to be valid, these instruments must be both appropriate and accurate in order to ensure the quality of the results.

Ageing in women has a significant impact on genital health, giving rise to a set of symptoms and signs collectively referred to as the genitourinary syndrome of menopause (GSM).

This clinical condition affects approximately 50% of postmenopausal women. While the urinary component of GSM can be quantified through validated diagnostic tests, vulvovaginal atrophy cannot be objectively measured. Its severity increases with advancing age, impacting self-esteem, well-being, and sexuality. Nevertheless, it often remains a taboo subject-stigmatized by women and under recognized by physicians. In this context, the DIVA questionnaire (Day-to-Day Impact of Vaginal Aging) combines the advantages of being practical for use in population-based studies, of transforming subjective measures into objective, quantifiable and analyzable data, and of assessing the relative weight of each domain or component of female genital atrophy on quality of life.

Other advantages of this questionnaire lie in the fact that it is a well-studied and validated instrument, with the ability to assess therapeutic interventions. It has also been adapted into languages other than English-including Spanish, Italian, German and Turkish-and has been validated within these cultural contexts.

The DIVA questionnaire assesses and quantifies the impact of female genital ageing. It consists of 23 items organised into four constructs, covering the following dimensions: daily activities, emotional well-being, sexual function, and self-concept/body image. Two versions of the questionnaire are available: the full version with 23 items, which includes four items within the sexual function construct that can only be answered by women who are sexually active; and a shorter version with 19 items, which can be applied regardless of sexual activity status. Each item is rated on a five-point Likert scale, and the score for each dimension is calculated as the mean of the corresponding items, with higher scores indicating a greater adverse impact of atrophic symptoms.

The inclusion criteria were assured by several filter questions, including at least one genital (vagina or vulvar) complain; symptoms such as 1-dryness, 2-irritation, 3-pruritus,4- burning or vaginal pain or after intercourse, 5- soreness or after intercourse, 6- dyspareunia, 7- bleed or bad smell discharge after sexual intercourse or other sexual activity.

A paper-pencil version of the survey was given to women participating at the screening trial, by one of our research partners.

The study was approved by the Ethical Commission for Health of Regional Health Administration of Lisbon and Tagus Valley (CES ARS-LVT) and the Ethical Commission of Local Health Unit of the Leiria Region.

For the normative convenience sample of the general population, participants will be recruited from a large urban primary care centre, the Sete Rios Personalized Health Care Unit (UCSP), in Lisbon. For the clinical convenience sample, participants will be recruited from the general gynecology outpatient clinic of a private hospital (Hospital Dom Manuel de Aguiar) and from the urogynecology outpatient clinic of a public hospital (Hospital Santo André), both located in an urban centre in Leiria.

The participants sample size was determined considering the recommendations of Hair et al. That is, dimension more than 100 participants and the rule of thumb has been at least 10 participants for each scale item, i.e., an ideal ratio of respondents to items is 10:18, corresponding to 23x10 that is at least 230.

The study variables are collected through a self-administered form completed by the participants. This form includes five questionnaires: a genital atrophy symptom questionnaire, sociodemographic data, the DIVA questionnaire, the EQ-5D, and the short version of the Female Sexual Function Questionnaire.

Recruitment for the project will be carried out by the investigators involved. Participant selection will be voluntary and conducted by convenience sampling, in a non-random manner. In all cases, individuals referred to the study must provide prior free and informed consent by signing the informed consent form, after confirmation that they meet all inclusion criteria and none of the exclusion criteria.

The participant will then be provided with the informed consent form to read carefully, while the study is explained orally. After obtaining written informed consent, the participant will complete the designated questionnaire form, identified by a participant ID number assigned sequentially. An investigator will always be available to clarify any questions that may arise during the self-completion of the form.

To evaluate psychometric properties of the questionnaire six measures will be addressed, namely:

Rate of completion and distribution of scores, structural validity with confirmatory factor analysis, assessment of internal consistency, inter- item and item-total correlation finally convergent and divergent validity. To this end, the data were entered and analysed in the Jamovi program.

ELIGIBILITY:
Inclusion Criteria:To present at least one symptom related to genital atrophy, referring to the external genitalia (vulva or vagina):

* dryness
* itching
* irritation
* discomfort on urination or during intercourse
* pain on urination or during intercourse
* bleeding during intercourse

Exclusion Criteria:

* pregnancy
* active cancer
* inability to speak Portuguese
* mental or physical condition that prevents providing coherent responses to the questionnaire.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women attending a medical consultation will be eligible for inclusion.
Study Population: Women attending a medical consultation will be eligible for inclusion. The normative convenience sample from the general population will be recruited from the south of Portugal, from a large urban primary care center, the Sete Rios Personalized Health Care Unit (UCSP), in Lisbon. The clinical convenience sample will be recruited from the general gynecology outpatient clinic of a private hospital (Hospital Dom Manuel de Aguiar) and from the urogynecology outpatient clinic of a public hospital (Hospital Santo André), both located in an urban center in Leiria. Also from the north of country recruitment will take place at a private clinical in Braga city.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Psychometric validation of Day to Day Impact of Vaginal Ageing Questionnaire (DIVA) to Portuguese Woman from Portugal Country. The methodological approach is a descriptive cross-sectional study of qualitative and quantitative variables. | Each patient complete the five questionnaires at baseline and a subset of 50 patients were selected to repeat the DIVA questionnaire and the Symptoms questionnaire 2 to 30 days after baseline to access Test-retest reliability.
  Primary outcome measure focuses on the psychometric validation of the portuguese version of the Day-to-Day Impact of Vaginal Aging (DIVA) questionnaire, including the evaluation of its internal consistency, factorial structure, construct validity, and test-retest reliability.
  The DIVA assesses the impact of vaginal aging symptoms in the daily activities, sexual function, emotional well-being, and self-concept/body image domains, with scores ranging from 0 to 92 (higher scores = worse impact).
  Two versions of the questionnaire are available: the full version with 23 items, which includes four items within the sexual function construct that can only be answered by women who are sexually active; and a shorter version with 19 items, which can be applied regardless of sexual activity status. Each item is rated on a five-point Likert scale, and the score for each dimension is calculated as the Mean of the corresponding items.

SECONDARY OUTCOMES:
Psychometric validation of Day to Day Impact of Vaginal Aging Questionnaire to Portuguese Woman with confirmatory factor analyses with other constructs | Each patient complete the five questionnaires at baseline and a subset of 50 patients were selected to repeat the DIVA questionnaire and the Symptoms questionnaire 2 to 30 days after baseline to access Test-retest reliability.
  Additional evidence of construct validity was obtained via examination of correlation with other measures of related constructs, such as Symptom Severity Questionnaire (assess the severity of symptoms related to vaginal atrophy: dryness, itching, burning, irritation, urinary pain, or pain/bleeding during intercourse) rated on a 5-point Likert scale (0 = no discomfort; 4 = extreme discomfort) the EuroQol 5D scale assesses general health-related quality of life across 5 domains, with scores ranging from 1 to 5, where higher scores indicate worse health outcomes. and Female Sexual Function Index -short form 6, assesses various domains of female sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. The total score ranges from 2 to 30, with higher scores indicating better sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia A Antunes, PhD Student, Principal Investigator — Minho University
Locations (1):
- Personalized Health Care Unit of Sete Rios, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No
Although the database is encrypted and does not contain personally identifiable elements, it contains a large amount of sensitive personal information that could generate inferences based on the location of origin where the questionnaire was collected.

REFERENCES:
- [Background] Santos Pechorro P, Monteiro Pascoal P, Monteiro Pereira N, Poiares C, Neves Jesus S, Xavier Vieira R. Validação da versão portuguesa do Índice de Funcionamento Sexual Feminino - 6. Published online 2016. doi:10.1016/j.androl.2016.06.001
- [Background] Ferreira PL, Ferreira LN, Pereira LN. [Contribution for the validation of the Portuguese version of EQ-5D]. Acta Med Port. 2013 Nov-Dec;26(6):664-75. Epub 2013 Dec 20. Portuguese. PMID 24388252
- [Background] Mokkink Cecilia AC Prinsen Donald L Patrick Jordi Alonso Lex M Bouter LB, Mokkink CL. COSMIN Study Design checklist for Patient-reported outcome measurement instruments. Accessed May 15, 2022. www.cosmin.nl
- [Background] Sert B, Ozgul S. Turkish day-to-day impact of vaginal aging questionnaire: reliability, validity and relationship with pelvic floor distress. Int Urogynecol J. 2022 Nov;33(11):3093-3102. doi: 10.1007/s00192-022-05085-w. Epub 2022 Jan 27. PMID 35084513
- [Background] Gabes M, Stute P, Apfelbacher C. Validation of the German Day-to-Day Impact of Vaginal Aging (DIVA) Questionnaire in Peri- and Postmenopausal Women. Sex Med. 2021 Aug;9(4):100382. doi: 10.1016/j.esxm.2021.100382. Epub 2021 Jun 12. PMID 34130226
- [Background] Moral E, Delgado JL, Carmona F, Caballero B, Guillan C, Gonzalez PM, Suarez-Almarza J, Velasco-Ortega S, Nieto Magro C; writing group of GENISSE study. The impact of genitourinary syndrome of menopause on well-being, functioning, and quality of life in postmenopausal women. Menopause. 2018 Dec;25(12):1418-1423. doi: 10.1097/GME.0000000000001148. PMID 29944636
- [Background] Hunter MM, Guthrie KA, Larson JC, Reed SD, Mitchell CM, Diem SJ, LaCroix AZ, Huang AJ. Convergent-Divergent Validity and Correlates of the Day-to-Day Impact of Vaginal Aging Domain Scales in the MsFLASH Vaginal Health Trial. J Sex Med. 2020 Jan;17(1):117-125. doi: 10.1016/j.jsxm.2019.10.010. Epub 2019 Dec 4. PMID 31812686
- [Background] Gabes M, Knuttel H, Stute P, Apfelbacher CJ. Measurement properties of patient-reported outcome measures (PROMs) for women with genitourinary syndrome of menopause: a systematic review. Menopause. 2019 Nov;26(11):1342-1353. doi: 10.1097/GME.0000000000001390. PMID 31688581
- [Background] Huang AJ, Gregorich SE, Kuppermann M, Nakagawa S, Van Den Eeden SK, Brown JS, Richter HE, Walter LC, Thom D, Stewart AL. Day-to-Day Impact of Vaginal Aging questionnaire: a multidimensional measure of the impact of vaginal symptoms on functioning and well-being in postmenopausal women. Menopause. 2015 Feb;22(2):144-54. doi: 10.1097/GME.0000000000000281. PMID 24983271
- [Background] Nappi RE, Palacios S, Panay N, Particco M, Krychman ML. Vulvar and vaginal atrophy in four European countries: evidence from the European REVIVE Survey. Climacteric. 2016 Apr;19(2):188-97. doi: 10.3109/13697137.2015.1107039. Epub 2015 Nov 19. PMID 26581580
- [Background] Nappi RE, Palacios S, Bruyniks N, Particco M, Panay N; EVES Study investigators. The burden of vulvovaginal atrophy on women's daily living: implications on quality of life from a face-to-face real-life survey. Menopause. 2019 May;26(5):485-491. doi: 10.1097/GME.0000000000001260. PMID 30422932
- [Background] Eremenco S, Pease S, Mann S, Berry P; PRO Consortium's Process Subcommittee. Patient-Reported Outcome (PRO) Consortium translation process: consensus development of updated best practices. J Patient Rep Outcomes. 2017;2(1):12. doi: 10.1186/s41687-018-0037-6. Epub 2018 Feb 27. PMID 29757299
- [Background] Calvert M, King M, Mercieca-Bebber R, Aiyegbusi O, Kyte D, Slade A, Chan AW, Basch E, Bell J, Bennett A, Bhatnagar V, Blazeby J, Bottomley A, Brown J, Brundage M, Campbell L, Cappelleri JC, Draper H, Dueck AC, Ells C, Frank L, Golub RM, Griebsch I, Haywood K, Hunn A, King-Kallimanis B, Martin L, Mitchell S, Morel T, Nelson L, Norquist J, O'Connor D, Palmer M, Patrick D, Price G, Regnault A, Retzer A, Revicki D, Scott J, Stephens R, Turner G, Valakas A, Velikova G, von Hildebrand M, Walker A, Wenzel L. SPIRIT-PRO Extension explanation and elaboration: guidelines for inclusion of patient-reported outcomes in protocols of clinical trials. BMJ Open. 2021 Jun 30;11(6):e045105. doi: 10.1136/bmjopen-2020-045105. PMID 34193486
- [Background] Mattos S, Moreira T, Pereira D, et al. INSTRUMENTS FOR MEASURING SELF-PERCEPTED HEALTH AMONG ADULTS: A SCOPING REVIEW. Psicol Saúde Doença. 2020;21(03):878- 895. doi:10.15309/20PSD210328

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT07250490/Prot_ICF_000.pdf